CLINICAL TRIAL: NCT04181762
Title: A Two-year, Phase III Randomized, Double-blind, Parallel-group, Placebo-controlled Trial to Evaluate the Safety, Efficacy, and Tolerability of 300 mg s.c. Secukinumab Versus Placebo, in Combination With SoC Therapy, in Patients With Active Lupus Nephritis
Brief Title: Study of Safety, Efficacy and Tolerability of Secukinumab Versus Placebo, in Combination With SoC Therapy, in Patients With Active Lupus Nephritis
Acronym: SELUNE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study terminated by sponsor due to futility analysis
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAIN457Q12301; 2019-003211-57 (EudraCT Number); PACTR202211748997845 (Other: PACTR)
Record Dates: First submitted 2019-11-27; First posted 2019-11-29 (Actual); Results first posted 2024-10-10 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Lupus Nephritis
Keywords: Systemic Lupus Erythematosus (SLE); Lupus Nephritis (LN); secukinumab; renal biopsy; estimated Glomerular Filtration Rate (eGFR); Urine Protein-to-Creatinine Ratio (UPCR); Standard of Care (SoC) background therapy
MeSH Terms: conditions — Lupus Nephritis; Lupus Erythematosus, Systemic | interventions — secukinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- secukinumab (Experimental): A blinded, weekly, subcutaneous (s.c.) secukinumab 300 mg loading regimen was administered for the first 4 weeks followed by a monthly maintenance dose in all randomized subjects thereafter.
  Interventions: Drug: secukinumab
- placebo (Placebo Comparator): A blinded, weekly, subcutaneous (s.c.) matching placebo loading regimen was administered for the first 4 weeks followed by a monthly maintenance dose in all randomized subjects thereafter.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: secukinumab — STUDY DRUG
  Other Names: AIN457
  Arms: secukinumab
Drug: Placebo — Placebo
  Arms: placebo

SUMMARY:
This was a pivotal, randomized, double-blind, placebo-controlled trial evaluating at Week 52 the efficacy and safety of secukinumab versus placebo in patients with active lupus nephritis (ISN/RPS Class III or IV, with or without co-existing class V features) also receiving background standard of care therapy (SoC).

DETAILED DESCRIPTION:
The study consisted of the following parts:

* Screening (up to 42 days/6 weeks)
* Run-in period (optional): For subjects who received Mycophenolic acid (MPA) as SoC induction therapy as per investigator's decision and who were not already on MPA at Screening, MPA dosing was initiated during a run-in period before Randomization (for up to 4 weeks prior to the first dose of secukinumab)
* Treatment Period: Duration of 104 weeks of treatment with secukinumab/placebo in addition to SoC treatment (with last dose given at Week 100)
* Secukinumab dosing was started with initial dosing of 300 mg s.c. injections at Baseline, Weeks 1, 2, 3, and 4, followed by dosing every 4 weeks
* Follow-up period: Duration of 8 weeks (last visit performed 12 weeks after last dose of study medication) for all except for subjects entering extension study CAIN457Q12301E1 (NCT05232864).

A total of 275 subjects were enrolled and were randomized to secukinumab 300 mg (n = 137) or placebo (n = 138) until study termination. Recruitment in this study was stopped on 26-May-2023. The CAIN457Q12301 study was terminated early by Novartis due to futile results from interim analysis 1 (IA1). There was no safety related reasons for early termination or concerns for the subjects in the study. The decision was made to terminate both the core and the related extension study in view of treatment futility of the core study.

ELIGIBILITY:
Key inclusion criteria:

1. Adult male and female subjects aged 18 - 75 years old at the time of Baseline.
2. Confirmed diagnosis of:

   * SLE with documented history of at least 4 of the 11 criteria for SLE as defined by the American College of Rheumatology (ACR) (Tan et al 1982) revised by (Hochberg 1997). [NOTE: The 4 criteria did not have to be present at the time of Screening], OR
   * LN as the sole clinical criterion in the presence of ANA or anti-dsDNA antibodies.
3. Active lupus nephritis, as defined by meeting the 4 following criteria:

   * Biopsy within 6 months prior to Screening visit indicating active glomerulonephritis WHO or ISN/RPS Class III or IV LN [excluding III (C), IV-S (C) and IV-G (C)]; patients are permitted to have co-existing Class V. If no biopsy was performed within 6 months of screening, a biopsy was to be performed during the Screening period
   * UPCR ≥ 1 mg/mg at Screening.
   * eGFR > 30 mL/min/1.73 m2 by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI).
   * Active urinary sediment (presence of cellular casts (RBC or WBC casts)) or hematuria (> 5 RBC per high power field or above the laboratory reference range).
4. Subjects must have currently been on MPA, or willing to initiate SoC induction therapy for LN according to the institutional practices using MPA or low-dose CYC in addition to corticosteroids. For guidance, see published guidelines such as by (Bertsias et al 2012, Hahn et al 2012).
5. Subjects must had been treated with anti-malarials (e.g. hydroxychloroquine), unless contra-indicated, and the dose had been stable for at least 10 days prior to Randomization.
6. Able to provide signed informed consent.

Key Exclusion criteria:

1. Severe renal impairment as defined by i.) Stage 4 CKD, or ii.) presence of oliguria (defined as a documented urine volume < 400 mL/24 h), or iii.) ESRD required dialysis or transplantation.
2. Known intolerance/hypersensitivity to MPA, or oral corticosteroids, or any component of the study drug(s).
3. Subjects received any other biologic immunomodulatory therapy within 6 months prior to Screening, excluding belimumab where 3 months were acceptable.
4. Previous exposure to secukinumab (AIN457) or any other biologic drug targeting IL-17 or the IL-17 receptor.
5. Subjects received any investigational drug within 1 month or five times the half-life of enrollment, whichever was longer.
6. Receipt of more than 3000 mg i.v. pulse methylprednisolone (cumulative dose) within the 12 weeks prior to Baseline.
7. Treatment with a systemic calcineurin inhibitor (e.g. cyclosporine, tacrolimus) within 12 weeks prior to Baseline
8. CYC use (i.v. or oral) within the month prior to Baseline.
9. Subjects requiring dialysis within the previous 12 months before Screening.
10. History of renal transplant.
11. Any severe progressive or uncontrolled concurrent medical condition, including recent severe thromboembolic events, that, in the opinion of the principal investigator, renders the subject unsuitable for the trial.
12. Active ongoing inflammatory diseases that might confound the evaluation of the benefit of secukinumab therapy, including inflammatory bowel disease.
13. Presence of investigator-identified significant medical problems which at the investigator's discretion would prevent the subject from participating in the study, included but not limited to the following: myocarditis, pericarditis, poorly controlled seizure disorder, acute confusional state, depression, severe manifestations of neuropsychiatric SLE (NPSLE).
14. Chest X-ray, computerized tomography (CT) scan, or MRI with evidence of ongoing infectious or malignant process, obtained within 3 months preceding the Screening visit and evaluated by a qualified physician.
15. History of chronic, recurrent systemic infections, active tuberculosis infection, or active systemic infections during the last two weeks (exception: common cold) prior to Randomization.
16. Known infection with human immunodeficiency virus (HIV), hepatitis B or hepatitis C at Screening or Randomization.
17. History of lymphoproliferative disease or any known malignancy or history of malignancy of any organ system treated or untreated within the past 5 years, regardless of whether there was evidence of local recurrence or metastases (except for skin Bowen's disease or basal cell carcinoma or actinic keratoses that had been treated with no evidence of recurrence in the past 12 weeks, carcinoma in situ of the cervix or non-invasive malignant colon polyps that had been removed).
18. Any of the following abnormal laboratory values on Screening evaluations as reported by Central Laboratory:

    * Aspartate aminotransferase (AST), alanine aminotransferase (ALT), or amylase > 2.5xULN
    * Hemoglobin < 8g/dL
    * Neutrophils < 1.0 x 109/L
    * Platelet count < 50 x 109/L

21. Pregnant or lactating women. 22. Women of childbearing potential, defined as all women physiologically capable of becoming pregnant, unless they were using highly effective methods of contraception during the entire study or longer if required by locally approved prescribing information (e.g., in European Union (EU) 20 weeks). Of note: the highly effective methods of contraception were mandated due to SoC medications used as per protocol (MPA and CYC).

In case local regulations deviated from the contraception methods listed above, local regulations applied and were described in the informed consent form (ICF).

If stricter female or male contraception requirements were specified in the country-specific label for induction and maintenance standard of care medications, they had to be followed.

Note: Women were considered post-menopausal and not of childbearing potential if they had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g., age appropriate, history of vasomotor symptoms) or had surgical bilateral oophorectomy (with or without hysterectomy), total hysterectomy or tubal ligation at least six weeks prior to enrollment. In the case of oophorectomy alone, only when the reproductive status of the woman had been confirmed by follow-up hormone level assessment was she considered not of childbearing potential.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Actual)
Dates: Start 2020-07-07 (Actual); Primary Completion 2023-09-13 (Actual); Study Completion 2023-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (93):
- United States (8):
  - University Of Alabama, Birmingham, Alabama
  - Kaiser Permanente Fontana, Fontana, California
  - University of California LA, Los Angeles, California
  - Arthritis and Rheum Dise Spec, Aventura, Florida
  - Integral Rheumatology and Immunology Specialists IRIS, Plantation, Florida
  - Piedmont Heart Institute, Atlanta, Georgia
  - Beth Israel Deaconess Hospital, Boston, Massachusetts
  - Ahmed Arif Medical Research Center, Grand Blanc, Michigan
- Argentina (3):
  - Novartis Investigative Site, Caba, Buenos Aires
  - Novartis Investigative Site, Ciudad Autonoma de Bs As, Buenos Aires
  - Novartis Investigative Site, Córdoba
- Novartis Investigative Site, Westmead, New South Wales, Australia
- Brazil (6):
  - Novartis Investigative Site, Fortaleza, Ceará
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, Joinville, Santa Catarina
  - Novartis Investigative Site, Santo André, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
  - Novartis Investigative Site, São José do Rio Preto
- Novartis Investigative Site, Toronto, Ontario, Canada
- Chile (4):
  - Novartis Investigative Site, Valdivia, Los Ríos Region
  - Novartis Investigative Site, Santiago, RM
  - Novartis Investigative Site, Concepción
  - Novartis Investigative Site, Santiago
- China (11):
  - Novartis Investigative Site, Nanning, Guangxi
  - Novartis Investigative Site, Shijiazhuang, Hebei
  - Novartis Investigative Site, Changsha, Hunan
  - Novartis Investigative Site, Nanchang, Jiangxi
  - Novartis Investigative Site, Binzhou, Shandong
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Chongqing
  - Novartis Investigative Site, Guangzhou
  - Novartis Investigative Site, Shanghai
  - Novartis Investigative Site, Wuhan
- Colombia (4):
  - Novartis Investigative Site, Medellín, Antioquia
  - Novartis Investigative Site, Barranquilla
  - Novartis Investigative Site, Cali
  - Novartis Investigative Site, Cundinamarca
- Novartis Investigative Site, Zagreb, Croatia
- Novartis Investigative Site, Prague, Czechia
- Novartis Investigative Site, Odense C, Denmark
- Novartis Investigative Site, Marseille, France
- Novartis Investigative Site, Mainz, Germany
- Greece (2):
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Thessaloniki
- Guatemala (2):
  - Novartis Investigative Site, Guatemala City
  - Novartis Investigative Site, Quetzaltenango
- Novartis Investigative Site, New Delhi, National Capital Territory of Delhi, India
- Novartis Investigative Site, Padua, PD, Italy
- Japan (5):
  - Novartis Investigative Site, Toyoake, Aichi-ken
  - Novartis Investigative Site, Kitakyushu, Fukuoka
  - Novartis Investigative Site, Sendai, Miyagi
  - Novartis Investigative Site, Kurashiki, Okayama-ken
  - Novartis Investigative Site, Chūō, Yamanashi
- Mexico (4):
  - Novartis Investigative Site, Mexicali, Baja California Norte
  - Novartis Investigative Site, Mexico City, Mexico CP
  - Novartis Investigative Site, Mérida, Yucatán
  - Novartis Investigative Site, México
- Novartis Investigative Site, Oslo, Norway
- Novartis Investigative Site, Santiago de Surco, Lima region, Peru
- Philippines (4):
  - Novartis Investigative Site, Lipa City, Batangas
  - Novartis Investigative Site, Iloilo City
  - Novartis Investigative Site, Manila
  - Novartis Investigative Site, Quezon
- Portugal (4):
  - Novartis Investigative Site, Coimbra
  - Novartis Investigative Site, Guimarães
  - Novartis Investigative Site, Lisbon
  - Novartis Investigative Site, Porto
- Romania (3):
  - Novartis Investigative Site, Oradea, Jud Bihor
  - Novartis Investigative Site, Râmnicu Vâlcea, Vâlcea County
  - Novartis Investigative Site, Bucharest
- Russia (5):
  - Novartis Investigative Site, Kazan'
  - Novartis Investigative Site, Kemerovo
  - Novartis Investigative Site, Rostov-on-Don
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Yaroslavl
- Novartis Investigative Site, Piešťany, Slovakia
- South Korea (2):
  - Novartis Investigative Site, Seoul, Seocho Gu
  - Novartis Investigative Site, Seoul
- Spain (3):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Santiago de Compostela, Galicia
  - Novartis Investigative Site, Vigo, Pontevedra
- Novartis Investigative Site, Stockholm, Sweden
- Novartis Investigative Site, Sankt Gallen, Switzerland
- Taiwan (3):
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Taoyuan District
- Novartis Investigative Site, Bangkok, Thailand
- Turkey (Türkiye) (2):
  - Novartis Investigative Site, Bakırkoy Istanbul
  - Novartis Investigative Site, Istanbul
- Vietnam (3):
  - Novartis Investigative Site, Ho Chi Minh City, VNM
  - Novartis Investigative Site, Hanoi
  - Novartis Investigative Site, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing access to patient-level data and supporting clinical documents from eligible studies with qualified external researchers. Requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to protect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Zhao MH, Cons Molina F, Aroca G, Tektonidou MG, Mathur A, Tangadpalli R, Sun R, Martin R, Pellet P, Ngoc Phuong Huynh T. Secukinumab in active lupus nephritis: Results from phase III, randomised, placebo-controlled study (SELUNE) and open-label extension study. Rheumatology (Oxford). 2025 Oct 15:keaf536. doi: 10.1093/rheumatology/keaf536. Online ahead of print. PMID 41092316
- [Derived] Avasare R, Drexler Y, Caster DJ, Mitrofanova A, Jefferson JA. Management of Lupus Nephritis: New Treatments and Updated Guidelines. Kidney360. 2023 Oct 1;4(10):1503-1511. doi: 10.34067/KID.0000000000000230. PMID 37528520
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2291

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in 106 centers in 34 countries worldwide.
Pre-assignment Details: At Baseline, all eligible subjects were randomized in a 1:1 ratio to secukinumab 300 mg s.c. or placebo via Interactive Response Technology (IRT).
Groups:
- Secukinumab 300 mg: A blinded, weekly, subcutaneous (s.c.) secukinumab 300 mg loading regimen was administered for the first 4 weeks followed by a monthly maintenance dose in all randomized subjects thereafter (maximum treatment exposure during the core study: 786 days).
- Placebo: A blinded, weekly, subcutaneous (s.c.) matching placebo loading regimen was administered for the first 4 weeks followed by a monthly maintenance dose in all randomized subjects thereafter (maximum treatment exposure during the core study: 794 days).
Period: Overall Study
Arm/Group | Secukinumab 300 mg | Placebo
Started (All randomized subjects were included in the Full Analysis Set and Safety Set.) | 137 | 138
Full Analysis Set 2 (All analyzable subjects from the randomized set to whom study treatment was assigned and who had or would have had an opportunity to reach 52 weeks of treatment at the study termination (including subjects who discontinued study treatment).) | 91 | 91
Pharmacokinetic Set (All subjects who had at least one PK/PD assessment and received at least one dose of study drug) | 136 | 0
Completed (Completed study) | 23 | 23
Not Completed | 114 | 115
Not completed — Adverse Event | 1 | 3
Not completed — Lost to Follow-up | 1 | 1
Not completed — Physician Decision | 1 | 3
Not completed — Pregnancy | 0 | 1
Not completed — Lack of Efficacy | 2 | 2
Not completed — Study terminated by sponsor | 95 | 97
Not completed — Subject decision | 11 | 4
Not completed — Death | 1 | 1
Not completed — Protocol deviation | 1 | 0
Not completed — Withdrawal of informed consent | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Secukinumab 300 mg | Placebo | Total
Number analyzed (Participants) | 137 | 138 | 275
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.1 (10.84) | 33.2 (11.28) | 33.6 (11.05)
Age, Customized [Count of Participants; unit: Participants]
  < 30 years | 55 | 64 | 119
  >= 30 years | 82 | 74 | 156
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 116 | 124 | 240
  Male | 21 | 14 | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 21 | 21 | 42
  Asian | 67 | 56 | 123
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 9 | 15
  White | 42 | 52 | 94
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Complete Renal Response (CRR) at Week 52
Description: Complete Renal Response (CRR) is a composite endpoint defined as:
  * Estimated Glomerular Filtration Rate (eGFR) >= 60 mL/min/1.73 m^2 or no less than 85% of core Baseline values and
  * 24-hour Urine-to-Protein Creatinine Ratio (UPCR) =< 0.5mg/mg
  * No treatment discontinuation before Week 52
  * The subject did not receive more than 10 mg/day prednisone or equivalent for >= 3 consecutive days or for >= 7 days in total during Week 44 through Week 52.
  Non-responder imputation (NRI) was used for participants who did not have the required data to compute responses at Week 52 or who had discontinued study treatment before Week 52. A logistic regression model was used for the analysis of this endpoint.
Time Frame: Baseline, Week 52
Population: Full Analysis Set 2.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Secukinumab 300 mg | Placebo
Number analyzed (Participants) | 91 | 91
Percentage of participants | 25.9 [16.8 to 34.9] | 38.6 [28.5 to 48.7]
Statistical Analysis 1: Comparison: Secukinumab 300 mg vs Placebo; Complete Renal Response (CRR) at Week 52; Test type: Superiority; p = 0.0662, Regression, Logistic; Mean Difference (Final Values) = -12.7, 95% CI 2-sided [-26.3 to 0.9] — Difference from placebo and 95% CI are from a logistic regression model with treatment group, stratification factor (SoC) and race as factors and baseline UPCR as a covariate using marginal standardization method

2. Secondary Outcome: Change From Baseline in 24-hour Urine Protein-to Creatinine Ratio (UPCR)
Description: Urine Protein-to-Creatinine Ratio (UPCR) was determined by a central laboratory by dividing the protein concentration by the creatinine concentration as measured in the urine collected (24-hour urine collection sample).
Time Frame: Baseline, Week 52
Population: Full Analysis Set. Only participants with a value at both Baseline and post-baseline visit included.
Measure: Mean (Standard Deviation); unit: mg/mg
Arm/Group | Secukinumab 300 mg | Placebo
Number analyzed (Participants) | 67 | 63
mg/mg | -2.204 (3.5162) | -2.741 (5.9448)

3. Secondary Outcome: Percentage of Participants Achieving Partial Renal Response (PRR) at Week 52
Description: Partial Renal Response (PRR) is a composite endpoint defined as:
  * >= 50% reduction in 24-hour Urine-to-Protein Creatinine Ratio (UPCR) to sub-nephrotic levels (=< 3 mg/mg) and
  * Estimated Glomerular Filtration Rate (eGFR) >= 60 mL/min/1.73 m^2 or no less than 85% of Baseline
Time Frame: Baseline, Week 52
Population: Full Analysis Set. Only participants with a value at both Baseline and post-baseline visit included.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Secukinumab 300 mg | Placebo
Number analyzed (Participants) | 73 | 72
Percentage of participants | 56.2 [44.1 to 67.8] | 63.9 [51.7 to 74.9]
Statistical Analysis 1: Comparison: Secukinumab 300 mg vs Placebo; Partial Renal Response (PRR) at Week 52; Test type: Other; Mean Difference (Final Values) = -7.7, 95% CI 2-sided [-23.7 to 8.4] — 95% Confidence Intervals (CIs) are constructed using the exact binomial test

4. Secondary Outcome: Average Daily Dose of Oral Corticosteroids
Description: Average daily dose of oral corticosteroids doses was used to assess efficacy of secukinumab compared to placebo in the averaged daily dose of oral corticosteroids administered between Week 16 and Week 52.
Time Frame: Week 16 to Week 52
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: mg/day
Arm/Group | Secukinumab 300 mg | Placebo
Number analyzed (Participants) | 137 | 138
mg/day | 8.1243 (6.38329) | 7.4791 (5.61958)

5. Secondary Outcome: Percentage of Participants Achieving Partial Renal Response (PRR) at Week 24
Description: as for outcome 3
Time Frame: Baseline, Week 24
Population: Full Analysis Set. Only participants with a value at both Baseline and post-baseline visit included.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Secukinumab 300 mg | Placebo
Number analyzed (Participants) | 108 | 110
Percentage of participants | 52.8 [42.9 to 62.5] | 43.6 [34.2 to 53.4]

6. Secondary Outcome: Incidence Rate of Participants Achieving Complete Renal Response (CRR) up to Week 52
Description: Time to achieve Complete Renal Response (CRR) up to week 52 was evaluated by 4-week interval by using Kaplan-Meier estimates. Participants who did not achieve CRR were censored at the date of their last non-missing CRR result (including participants who completed week 52 without achieving CRR).
  * Subjects at risk = Subjects who did not achieve CRR and were not censored before or at the start of the specified interval. Participants had an event when achieving CRR.
  * Incidence rate (%) = (number of subjects with event/number of subjects at risk) x 100.
Time Frame: Baseline to Week 52
Population: Participants in the Full Analysis Set with an available value for the outcome measure. Day 1 = Date of randomization.
Measure: Number; unit: Percentage of participants
Arm/Group | Secukinumab 300 mg | Placebo
Number analyzed (Participants) | 131 | 132
Percentage of participants
  1 to 28 days | 0.0 | 0.8
  29 to 56 days: number analyzed (Participants) | 130 | 130
  29 to 56 days | 0.0 | 0.0
  57 to 84 days: number analyzed (Participants) | 129 | 130
  57 to 84 days | 3.1 | 5.4
  85 to 112 days: number analyzed (Participants) | 120 | 119
  85 to 112 days | 11.7 | 16.8
  113 to 140 days: number analyzed (Participants) | 103 | 91
  113 to 140 days | 0.0 | 2.2
  141 to 168 days: number analyzed (Participants) | 101 | 88
  141 to 168 days | 0.0 | 3.4
  169 to 196 days: number analyzed (Participants) | 98 | 80
  169 to 196 days | 20.4 | 20.0
  197 to 224 days: number analyzed (Participants) | 69 | 57
  197 to 224 days | 1.4 | 0.0
  225 to 252 days: number analyzed (Participants) | 65 | 56
  225 to 252 days | 0.0 | 0.0
  253 to 280 days: number analyzed (Participants) | 61 | 55
  253 to 280 days | 14.8 | 3.6
  281 to 308 days: number analyzed (Participants) | 46 | 47
  281 to 308 days | 0.0 | 2.1
  309 to 336 days: number analyzed (Participants) | 45 | 44
  309 to 336 days | 0.0 | 0.0
  337 to 364 days: number analyzed (Participants) | 43 | 41
  337 to 364 days | 2.3 | 7.3

7. Secondary Outcome: Incidence Rate of Participants Achieving Partial Renal Response (PRR) up to Week 52
Description: Time to achieve Partial Renal Response (PRR) up to week 52 was evaluated by 4-week interval by using Kaplan-Meier estimates. Participants who did not achieve PRR were censored at the date of their last non-missing PRR result (including participants who completed week 52 without achieving PRR). Participants had event when achieving PRR.
  * Subjects at risk = Subjects who did not achieve PRR and were not censored before or at the start of the specified interval.
  * Incidence rate (%) = (number of subjects with event/ number of subjects at risk) x 100.
Time Frame: Baseline to Week 52
Population: Participants in the Full Analysis Set with an available value for the outcome measure. Day 1 = Date of randomization.
Measure: Number; unit: Percentage of participants
Arm/Group | Secukinumab 300 mg | Placebo
Number analyzed (Participants) | 131 | 132
Percentage of participants
  1 to 28 days | 0.0 | 0.8
  29 to 56 days: number analyzed (Participants) | 130 | 130
  29 to 56 days | 0.0 | 0.0
  57 to 84 days: number analyzed (Participants) | 129 | 130
  57 to 84 days | 7.0 | 5.4
  85 to 112 days: number analyzed (Participants) | 115 | 118
  85 to 112 days | 27.8 | 30.5
  113 to 140 days: number analyzed (Participants) | 79 | 76
  113 to 140 days | 1.3 | 2.6
  141 to 168 days: number analyzed (Participants) | 77 | 74
  141 to 168 days | 0.0 | 4.1
  169 to 196 days: number analyzed (Participants) | 74 | 67
  169 to 196 days | 32.4 | 14.9
  197 to 224 days: number analyzed (Participants) | 41 | 52
  197 to 224 days | 2.4 | 0.0
  225 to 252 days: number analyzed (Participants) | 38 | 50
  225 to 252 days | 2.6 | 0.0
  253 to 280 days: number analyzed (Participants) | 34 | 49
  253 to 280 days | 11.8 | 16.3
  281 to 308 days: number analyzed (Participants) | 25 | 35
  281 to 308 days | 4.0 | 2.9
  309 to 336 days: number analyzed (Participants) | 24 | 34
  309 to 336 days | 0.0 | 0.0
  337 to 364 days: number analyzed (Participants) | 22 | 31
  337 to 364 days | 0.0 | 6.5

8. Secondary Outcome: Time to Achieve First Morning Void Urine Protein-to-Creatinine Ratio (UPCR) <= 0.5 mg/mg up to Week 52
Description: Time to achieve first morning void Urine Protein-to-Creatinine Ratio (UPCR) <= 0.5 mg/mg up to week 52 was evaluated by 4-week interval by using Kaplan-Meier estimates. Participants who did not achieve UCPR were censored at the date of their last non-missing UCPR result (including participants who completed week 52 without achieving UCPR). Participants had event when achieving UCPR.
  * Subjects at risk = Subjects who did not achieve UCPR and were not censored before or at the start of the specified interval.
  * Incidence rate (%) = (number of subjects with event/ number of subjects at risk) x 100.
Time Frame: Baseline to Week 52
Population: Participants in the Full Analysis Set with an available value for the outcome measure. Day 1 = Date of randomization.
Measure: Number; unit: Percentage of participants
Arm/Group | Secukinumab 300 mg | Placebo
Number analyzed (Participants) | 135 | 136
Percentage of participants
  1 to 28 days | 19.3 | 21.3
  29 to 56 days: number analyzed (Participants) | 108 | 107
  29 to 56 days | 2.8 | 5.6
  57 to 84 days: number analyzed (Participants) | 104 | 100
  57 to 84 days | 8.7 | 7.0
  85 to 112 days: number analyzed (Participants) | 93 | 93
  85 to 112 days | 11.8 | 9.7
  113 to 140 days: number analyzed (Participants) | 79 | 81
  113 to 140 days | 7.6 | 7.4
  141 to 168 days: number analyzed (Participants) | 71 | 72
  141 to 168 days | 9.9 | 6.9
  169 to 196 days: number analyzed (Participants) | 62 | 63
  169 to 196 days | 9.7 | 3.2
  197 to 224 days: number analyzed (Participants) | 53 | 59
  197 to 224 days | 7.5 | 11.9
  225 to 252 days: number analyzed (Participants) | 48 | 50
  225 to 252 days | 4.2 | 6.0
  253 to 280 days: number analyzed (Participants) | 45 | 45
  253 to 280 days | 4.4 | 0.0
  281 to 308 days: number analyzed (Participants) | 41 | 44
  281 to 308 days | 12.2 | 4.5
  309 to 336 days: number analyzed (Participants) | 36 | 39
  309 to 336 days | 0.0 | 5.1
  337 to 364 days: number analyzed (Participants) | 32 | 34
  337 to 364 days | 3.1 | 2.9

9. Secondary Outcome: Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-Fatigue) Mean Change From Baseline up to Week 52
Description: The FACIT-Fatigue is a 13-item questionnaire that assesses self-reported fatigue and its impact upon daily activities and function over the past week. The purpose of the FACIT-Fatigue in this study was to assess the impact of fatigue on subjects with lupus nephritis (LN). The level of fatigue was measured on a 5-point Likert scale (0 = not at all, 1 = a little bit, 2 = somewhat, 3 = quite a bit, 4 = very much) based on their experience of fatigue during the past 2 weeks. The scale score is computed by summing the item scores, after reversing those items that are worded in the negative direction. FACIT-Fatigue scale score range from 0 to 52, where higher scores represent less fatigue.
Time Frame: Baseline, Week 12, Week 24, Week 36, Week 52
Population: Full Analysis Set. Only participants with a value at both Baseline and post-baseline visit included.
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | Secukinumab 300 mg | Placebo
Number analyzed (Participants) | 131 | 131
Unit on a scale
  Week 12 | -2.8 (8.47) | -1.9 (8.46)
  Week 24: number analyzed (Participants) | 118 | 116
  Week 24 | -1.4 (9.66) | -2.0 (8.93)
  Week 36: number analyzed (Participants) | 99 | 93
  Week 36 | -2.6 (9.21) | -2.1 (9.67)
  Week 52: number analyzed (Participants) | 82 | 79
  Week 52 | -2.0 (10.18) | -2.0 (9.51)

10. Secondary Outcome: Short Form Health Survey (SF-36) Version 2 (Acute Form) Mean Change From Baseline in Physical Component Score (PCS) up to Week 52
Description: The SF-36 questionnaire consists of eight scales yielding two summary measures: physical and mental health. The physical health measure includes four scales of physical functioning (10 items), role-physical (4 items), bodily pain (2 items), and general health (5 items). The mental health measure is composed of vitality (4 items), social functioning (2 items), role-emotional (3 items), and mental health (5 items). In this trial, SF-36-PCS responder (improvement of >= 2.5 points) were evaluated. Responses to items allow for direct calculation of scale scores, while the physical component summary (PCS) scores are computed from weighted scale scores. For all scales and summary measures, higher scores indicate better health outcomes (PCS scores range 0 to 100).
Time Frame: Baseline, Week 12, Week 24, Week 36, Week 52
Population: Full Analysis Set. Only participants with a value at both Baseline and post-baseline visit included.
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | Secukinumab 300 mg | Placebo
Number analyzed (Participants) | 131 | 131
Unit on a scale
  Week 12 | 2.306 (6.4306) | 2.210 (6.8760)
  Week 24: number analyzed (Participants) | 118 | 116
  Week 24 | 2.873 (6.4502) | 1.687 (6.5346)
  Week 36: number analyzed (Participants) | 99 | 93
  Week 36 | 2.910 (6.8234) | 3.152 (7.0623)
  Week 52: number analyzed (Participants) | 82 | 79
  Week 52 | 3.410 (7.7123) | 2.707 (6.8887)

11. Secondary Outcome: Lupus Quality of Life (LupusQoL) Physical Health Score Mean Change From Baseline up to Week 52
Description: The LupusQoL is a disease-specific, 34-item, self-report questionnaire designed to measure the health-related quality of life (HRQoL) of subjects with SLE within 8 domains (i.e., physical health (8 items), emotional health (6 items), body image (5 items), pain (3 items), planning (3 items), fatigue (4 items), intimate relationships (2 items), and burden to others (3 items)). Responses are based on a 5-point Likert scale where 0 (all of the time) to 4 (never). Each domain of the LupusQoL was scored separately. Transformed scores range from 0 (worst HRQoL) to 100 (best HRQoL).
Time Frame: Baseline, Week 12, Week 24, Week 36, Week 52
Population: Full Analysis Set. Only participants with a value at both Baseline and post-baseline visit included.
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | Secukinumab 300 mg | Placebo
Number analyzed (Participants) | 131 | 131
Unit on a scale
  Week 12 | 5.32 (16.031) | 6.18 (19.248)
  Week 24: number analyzed (Participants) | 118 | 116
  Week 24 | 4.84 (18.184) | 5.55 (20.485)
  Week 36: number analyzed (Participants) | 99 | 93
  Week 36 | 5.59 (20.684) | 7.89 (23.112)
  Week 52: number analyzed (Participants) | 82 | 79
  Week 52 | 7.62 (23.275) | 8.55 (20.589)

12. Secondary Outcome: Incidence of Adverse Events (AEs), Serious Adverse Events (SAEs)
Description: The distribution of adverse events was done via the analysis of frequencies for treatment emergent Adverse Event (TEAEs), Serious Adverse Event (TESAEs) and Deaths due to AEs, through the monitoring of relevant clinical and laboratory safety parameters.
Time Frame: From first dose of study treatment up to approximately 2 years
Population: Safety Set (SAF).
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab 300 mg | Placebo
Number analyzed (Participants) | 137 | 138
Participants
  Deaths | 1 | 1
  Serious Adverse Event (TESAEs) | 30 | 39
  Treatment Emergent Adverse Event (TEAEs) | 120 | 123
  TESAEs leading to study medication discontinuation | 8 | 10

13. Secondary Outcome: Percentage of Participants With Complete Renal Response (CRR) at Week 104 Within Those Who Had Achieved CRR at Week 52 in the Secukinumab Group
Description: The percentage of participants with maintained renal response (CRR) at Week 104 in the secukinumab group was evaluated
Time Frame: Week 52 to Week 104
Population: Participants in the Full Analysis Set who received secukinumab. Subset of participants who achieved CRR at Week 52 and had an available CRR assessment at Week 104.
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab 300 mg
Number analyzed (Participants) | 6
Participants
  Achieve CRR | 5
  Not Achieve CRR | 1

14. Secondary Outcome: Percentage of Participants With Improved or Maintained Response (PRR or CRR) at Week 104 in Those Who Had Achieved at Least PRR at Week 52 in the Secukinumab Group
Description: The percentage of participants with improved or maintained renal response (CRR) at Week 104 in the secukinumab group was evaluated
Time Frame: Week 52 to Week 104
Population: Participants in the Full Analysis Set who received secukinumab. Subset of participants who achieved PRR or CRR at Week 52 and had an available PRR or CRR assessment at Week 104.
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab 300 mg
Number analyzed (Participants) | 12
Participants
  Achieve PRR or CRR | 11
  Not achieve PRR or CRR | 1

ADVERSE EVENTS:
Time Frame: On-treatment adverse events and deaths were reported from first dose of study treatment to 84 days after last dose of study medication, assessed up to approximately 2 years.
Description: Any sign or symptom that occurred during the treatment and safety follow-up. The Safety Set included all subjects who received at least one dose of study treatment.
Arm/Group | Secukinumab 300 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 1/137 | 1/138
Serious Adverse Events (participants affected / at risk) | 30/137 | 39/138
Other Adverse Events (participants affected / at risk) | 111/137 | 116/138
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Secukinumab 300 mg (N=137) | Placebo (N=138)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Blood loss anaemia (Blood and lymphatic system disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1
Cataract (Eye disorders) | 2 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 1
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Generalised oedema (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1
Anaphylactic reaction (Immune system disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1
Hypogammaglobulinaemia (Immune system disorders) | 0 | 1
COVID-19 (Infections and infestations) | 3 | 4
Cellulitis (Infections and infestations) | 0 | 1
Chronic sinusitis (Infections and infestations) | 0 | 1
Dengue fever (Infections and infestations) | 0 | 1
Dengue haemorrhagic fever (Infections and infestations) | 0 | 1
Diarrhoea infectious (Infections and infestations) | 1 | 0
Endometritis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 1
Genital herpes (Infections and infestations) | 0 | 1
Haematological infection (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Herpes zoster disseminated (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 0
Meningitis (Infections and infestations) | 1 | 0
Oesophageal candidiasis (Infections and infestations) | 1 | 0
Parotitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 5 | 3
Pneumonia bacterial (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 0
Pyelonephritis acute (Infections and infestations) | 2 | 1
Renal cyst infection (Infections and infestations) | 1 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 1 | 0
Soft tissue infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 2
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Hypervolaemia (Metabolism and nutrition disorders) | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 | 1
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 1
Dyskinesia (Nervous system disorders) | 0 | 1
Incoherent (Nervous system disorders) | 0 | 1
Intracranial pressure increased (Nervous system disorders) | 0 | 1
Post herpetic neuralgia (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Bipolar disorder (Psychiatric disorders) | 0 | 1
Major depression (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 4
Azotaemia (Renal and urinary disorders) | 0 | 1
End stage renal disease (Renal and urinary disorders) | 0 | 1
Lupus nephritis (Renal and urinary disorders) | 4 | 5
Nephrotic syndrome (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1
Endometriosis (Reproductive system and breast disorders) | 0 | 1
Genital tract inflammation (Reproductive system and breast disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
Hypertensive urgency (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Secukinumab 300 mg (N=137) | Placebo (N=138)
Anaemia (Blood and lymphatic system disorders) | 12 | 13
Iron deficiency anaemia (Blood and lymphatic system disorders) | 3 | 4
Leukopenia (Blood and lymphatic system disorders) | 6 | 10
Lymphopenia (Blood and lymphatic system disorders) | 3 | 1
Neutropenia (Blood and lymphatic system disorders) | 3 | 3
Dry eye (Eye disorders) | 3 | 2
Vision blurred (Eye disorders) | 3 | 6
Abdominal pain (Gastrointestinal disorders) | 3 | 6
Abdominal pain upper (Gastrointestinal disorders) | 2 | 4
Aphthous ulcer (Gastrointestinal disorders) | 3 | 2
Constipation (Gastrointestinal disorders) | 1 | 6
Diarrhoea (Gastrointestinal disorders) | 23 | 21
Dyspepsia (Gastrointestinal disorders) | 5 | 2
Gastritis (Gastrointestinal disorders) | 4 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 5
Haemorrhoids (Gastrointestinal disorders) | 3 | 1
Mouth ulceration (Gastrointestinal disorders) | 5 | 3
Nausea (Gastrointestinal disorders) | 11 | 5
Toothache (Gastrointestinal disorders) | 3 | 2
Vomiting (Gastrointestinal disorders) | 7 | 4
Chest discomfort (General disorders) | 3 | 0
Fatigue (General disorders) | 4 | 2
Oedema (General disorders) | 2 | 4
Oedema peripheral (General disorders) | 3 | 8
Peripheral swelling (General disorders) | 4 | 2
Pyrexia (General disorders) | 8 | 3
Bronchitis (Infections and infestations) | 3 | 3
COVID-19 (Infections and infestations) | 25 | 22
Conjunctivitis (Infections and infestations) | 1 | 4
Gastroenteritis (Infections and infestations) | 6 | 7
Herpes zoster (Infections and infestations) | 10 | 7
Influenza (Infections and infestations) | 3 | 3
Nasopharyngitis (Infections and infestations) | 11 | 11
Oral candidiasis (Infections and infestations) | 8 | 3
Oral herpes (Infections and infestations) | 5 | 2
Pharyngitis (Infections and infestations) | 4 | 11
Pneumonia (Infections and infestations) | 6 | 0
Upper respiratory tract infection (Infections and infestations) | 19 | 26
Urinary tract infection (Infections and infestations) | 19 | 30
Viral upper respiratory tract infection (Infections and infestations) | 1 | 3
Contusion (Injury, poisoning and procedural complications) | 2 | 4
Weight increased (Investigations) | 4 | 3
White blood cell count decreased (Investigations) | 2 | 3
Dyslipidaemia (Metabolism and nutrition disorders) | 7 | 5
Hypercholesterolaemia (Metabolism and nutrition disorders) | 3 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 4 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 7 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 9 | 11
Iron deficiency (Metabolism and nutrition disorders) | 1 | 3
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 | 19
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 4
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 | 4
Dizziness (Nervous system disorders) | 6 | 3
Headache (Nervous system disorders) | 21 | 14
Tremor (Nervous system disorders) | 3 | 2
Anxiety (Psychiatric disorders) | 3 | 4
Depression (Psychiatric disorders) | 3 | 2
Insomnia (Psychiatric disorders) | 8 | 6
Acute kidney injury (Renal and urinary disorders) | 6 | 2
Lupus nephritis (Renal and urinary disorders) | 2 | 3
Menstrual disorder (Reproductive system and breast disorders) | 6 | 1
Menstruation irregular (Reproductive system and breast disorders) | 4 | 1
Vaginal discharge (Reproductive system and breast disorders) | 1 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 14
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Acne (Skin and subcutaneous tissue disorders) | 1 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 6 | 11
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 3
Rash (Skin and subcutaneous tissue disorders) | 1 | 5
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 3
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 5 | 1
Hypertension (Vascular disorders) | 8 | 8
Hypotension (Vascular disorders) | 5 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2023-02-17): https://cdn.clinicaltrials.gov/large-docs/62/NCT04181762/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-09): https://cdn.clinicaltrials.gov/large-docs/62/NCT04181762/SAP_001.pdf